CLINICAL TRIAL: NCT02224495
Title: The Effect of Exercise Training on Cardiac Structure and Function
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gaia Hospital (Other)
Collaborators: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Ricardo Fontes Carvalho, MD, PhD, Gaia Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ET2011
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Standard of care
- Structured exercise training (Experimental): 8-week outpatient exercise-training program, encompassing 3 sessions per week, including endurance and resistance training
  Interventions: Behavioral: Structured exercise training

INTERVENTIONS:
Behavioral: Structured exercise training
  Arms: Structured exercise training

SUMMARY:
Exercise training, as part of cardiac rehabilitation, is effective in improving functional capacity and quality of life in patients with coronary artery disease. Other cardiovascular and non-cardiovascular benefits have been reported, namely in glucose metabolism, skeletal muscle function, oxidative stress, vascular function, pulmonary circulation, ischaemia-reperfusion lesion and ventricular remodelling.

However, the benefit of exercise training on systolic and diastolic function is controversial especially after acute myocardial infarction where no longitudinal study has evaluated diastolic function using modern echocardiographic parameters.

The hypothesis is that a structured program of exercise training can improve systolic and diastolic function in patients after myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Patients one month after myocardial infarction
* Older 18 years

Exclusion Criteria:

* Age above 75 years,
* Inability to exercise,
* Hemodinamically significant valvular disease,
* Moderate to severe chronic lung disease (vital capacity and/or forced expiratory volume in 1 s <80% of age-dependent predicted value),
* Atrial fibrillation
* Exercise induced myocardial ischemia
* Anaemia (haemoglobin <12 g/dl).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Myocardial early diastolic velocity at mitral annulus by tissue Doppler (E' velocity) | 4 months
  Determined by echocardiography; results in cm/s

SECONDARY OUTCOMES:
Ratio between early diastolic filling velocity from mitral inflow and myocardial early diastolic velocity at mitral annulus by tissue Doppler (E/E' ratio) | 4 months
  Determined by echocardiography; no unit (ratio)
Myocardial systolic velocity at mitral annulus by tissue Doppler (S' velocity) | 4 months
  Determined by echocardiography; results in cm/s
Left ventriclular ejection fraction | 4 months
  Determined by echocardiography; results in %

CONTACTS AND LOCATIONS:
Overall Officials: Adelino Leite-Moreira, PhD, Study Director — Universidade do Porto
Locations (1):
- Cardiology Department Gaia Hospital Center, Gaia, Portugal

REFERENCES:
- [Derived] Fontes-Carvalho R, Sampaio F, Teixeira M, Gama V, Leite-Moreira AF. The role of a structured exercise training program on cardiac structure and function after acute myocardial infarction: study protocol for a randomized controlled trial. Trials. 2015 Mar 12;16:90. doi: 10.1186/s13063-015-0612-6. PMID 25872588